CLINICAL TRIAL: NCT05097937
Title: Neurophysiological Effects of Percutaneous Electrolysis Related to Endogenous Pain Modulation
Brief Title: Analgesic Mechanisms of Percutaneous Electrolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Sergio Varela Rodríguez, PhD candidate, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EP550
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Percutaneous Electrolysis; Pain; Analgesia; Pain Modulation; Endogenous Analgesia System
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham intervention (Sham Comparator): The needle will be inserted for 90 seconds without galvanic current.
  Interventions: Other: Sham intervention
- Low intensity percutaneous electrolysis (Experimental): Galvanic current will be applied with an intensity of 0.3 mA for 90 seconds.
  Interventions: Other: Low intensity percutaneous electrolysis
- High intensity percutaneous electrolysis (Experimental): Participants will receive three impacts of galvanic current with an intensity of 3 mA for 3 seconds each.
  Interventions: Other: High intensity percutaneous electrolysis

INTERVENTIONS:
Other: Sham intervention — The needle will be inserted into the right common extensor tendon of the epicondyle for 90 seconds without galvanic current.
  Arms: Sham intervention
Other: Low intensity percutaneous electrolysis — A single impact of galvanic current will be applied in the common extensor tendon of the epicondyle (right side) with an intensity of 0.3 mA for 90 seconds.
  Arms: Low intensity percutaneous electrolysis
Other: High intensity percutaneous electrolysis — Three impacts of galvanic current will be applied in the common extensor tendon of the epicondyle (right side) with an intensity of 3 mA and a duration of 3 seconds each.
  Arms: High intensity percutaneous electrolysis

SUMMARY:
Percutaneous electrolysis is based on the application of a galvanic current through an acupuncture needle. The underlying mechanisms that explain the efficacy of this technique are not completely well understood. The objective is to delve into the neurophysiological analgesic effects of percutaneous electrolysis. Participants will be assigned to one of three intervention groups. The analgesic effects of the technique will be evaluated by means of variables related to endogenous pain modulation.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects
* Signature of the informed consent

Exclusion Criteria:

* Fear of needles
* Any pathology or process that causes pain
* Neurological, rheumatologic, cardiovascular or metabolic diseases
* Cutaneous alterations and cognitive or sensitivity disorders
* Pregnancy
* Recent intake of alcohol or caffeine
* Vigorous physical activity on the day of testing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Pressure Pain Thresholds (PPT) | Baseline and immediately after the intervention
  PPTs will be measure by algometry in the common extensor tendon of the epicondyle, bicipital groove and tibialis anterior muscle (all of the right side).

SECONDARY OUTCOMES:
Changes from baseline in Conditioned Pain Modulation (CPM) | Baseline and immediately after the intervention
  CPM will be assess by upper extremity submaximal effort tourniquet test with algometric measures in the common extensor tendon of the epicondyle, bicipital groove and tibialis anterior muscle (all of the right side).
Changes from baseline in Temporal Summation (TS) | Baseline and immediately after the intervention
  Assessed by Verbal Numeric Rating Scale (11-point). 10 consecutive pressures will be applied in the three previous locations (epicondyle, bicipital groove and tibialis anterior) with the algometer at the intensity of the pressure pain threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermería y Fisioterapia de la Universidad de Salamanca, Salamanca, Spain

REFERENCES:
- [Background] de Miguel Valtierra L, Salom Moreno J, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL. Ultrasound-Guided Application of Percutaneous Electrolysis as an Adjunct to Exercise and Manual Therapy for Subacromial Pain Syndrome: A Randomized Clinical Trial. J Pain. 2018 Oct;19(10):1201-1210. doi: 10.1016/j.jpain.2018.04.017. Epub 2018 May 16. PMID 29777953
- [Background] Garcia Bermejo P, De La Cruz Torres B, Naranjo Orellana J, Albornoz Cabello M. Autonomic Responses to Ultrasound-Guided Percutaneous Needle Electrolysis: Effect of Needle Puncture or Electrical Current? J Altern Complement Med. 2018 Jan;24(1):69-75. doi: 10.1089/acm.2016.0339. Epub 2017 Jan 30. PMID 28135129
- [Background] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Background] Abat F, Valles SL, Gelber PE, Polidori F, Stitik TP, Garcia-Herreros S, Monllau JC, Sanchez-Ibanez JM. [Molecular repair mechanisms using the Intratissue Percutaneous Electrolysis technique in patellar tendonitis]. Rev Esp Cir Ortop Traumatol. 2014 Jul-Aug;58(4):201-5. doi: 10.1016/j.recot.2014.01.002. Epub 2014 May 10. Spanish. PMID 24821478
- [Background] Abat F, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Clinical results after ultrasound-guided intratissue percutaneous electrolysis (EPI(R)) and eccentric exercise in the treatment of patellar tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1046-52. doi: 10.1007/s00167-014-2855-2. Epub 2014 Jan 30. PMID 24477495
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039